CLINICAL TRIAL: NCT01011439
Title: Phase II Study Of Oral PHA-848125AC In Patients With Thymic Carcinoma Previously Treated With Chemotherapy
Brief Title: Phase II Study Of Oral PHA-848125AC In Patients With Thymic Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: For the 2 last patients still on treated nominal therapeutic use of the Milciclib was approved at INT Milano.
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDKO-125a-006; 2009-014338-79 (EudraCT Number)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Thymic Carcinoma
Keywords: B3 and C malignant thymoma
MeSH Terms: conditions — Thymoma | interventions — N,1,4,4-tetramethyl-8-((4-(4-methylpiperazin-1-yl)phenyl)amino)-4,5-dihydro-1H-pyrazolo(4,3-h)quinazoline-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Milciclib Maleate (PHA-848125AC) (Experimental): 100 and 50 mg Capsule 150 mg/day once daily, for 7 consecutive days (days 1 to 7) followed by 7 days of rest (days 8 to 14) in a 2-week cycle
  Interventions: Drug: Milciclib Maleate

INTERVENTIONS:
Drug: Milciclib Maleate — 150 mg/day once daily, for 7 consecutive days (days 1 to 7) followed by 7 days of rest (days 8 to 14) in a 2-week cycle.
  Number of cycles: until disease progression or unacceptable toxicity.
  Other Names: PHA-848125AC

SUMMARY:
The intent of the study is to assess the antitumor activity of PHA-848125AC as second-line treatment in patients with recurrent or metastatic, unresectable thymic carcinoma previously treated with chemotherapy.

DETAILED DESCRIPTION:
The Simon's optimal 2 stage design is adopted for this single-arm, open-label, multicenter phase II clinical trial of PHA-848125AC administered to patients with recurrent or metastatic, unresectable thymic carcinoma previously treated with chemotherapy (only one prior systemic therapy allowed). The intent of the study is to assess the antitumor activity of PHA-848125AC and ultimately to improve the outcome of patients with thymic carcinoma who have already exploited one chemotherapy option. The primary end point for this study is a progression free survival rate of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of unresectable B3 thymoma or thymic carcinoma recurrent or progressing after prior chemotherapy (only one prior systemic therapy allowed)
* Presence of measurable disease
* Age >=18 years
* ECOG performance status 0-1
* Negative pregnancy test (if female in reproductive years)
* Use of effective contraceptive methods if men and women of child producing potential
* Adequate liver function Total Serum Bilirubin <=1.5 x upper limit of normal (ULN) Transaminases (AST/ALT) <=2.5ULN (if liver metastases are present, then <=5ULN is allowed) ALP <=2.5ULN (if liver and/or bone metastases are present, then <=5ULN is allowed)
* Adequate renal function Serum Creatinine <=ULN or Creatinine Clearance calculated by Cockcroft and Gault's formula > 60 mL/min.
* Adequate hematologic status ANC >=1,500cells/mm3 Platelet Count >=100,000cells/mm3 Hemoglobin >=9.0g/dL
* Two weeks must have elapsed since completion of prior chemotherapy, minor surgery, radiotherapy (provided that no more than 25% of bone marrow reserve has been irradiated)
* Resolution of all acute toxic effects of any prior treatments to NCI CTC (Version 3.0) grade <=1

Exclusion Criteria:

* Any of the following in the past 6 months: myocardial infarction, uncontrolled cardiac arrhythmia, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis
* Grade >1 retinopathy
* Known brain metastases
* Known active infections
* Pregnant or breast feeding women
* Diabetes mellitus uncontrolled
* Gastrointestinal disease that would impact on drug absorption
* Patients under treatment with anticoagulants or with coagulation disorders or with signs of hemorrhage at baseline
* Patients with previous history or current presence of neurological disorders, including epilepsy (although controlled by anticonvulsant therapy), Parkinson's disease and extra-pyramidal syndromes
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-02-22 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen Weiss, MD, Principal Investigator — Scottsdale Clinical Research Institute, USA; Benjamin Besse, MD, Principal Investigator — Institut Gustave Roussy, Villejuif, France; Julien Mazières, MD, Principal Investigator — Hopital Larrey CHU, Toulouse, France; Silvia Novello, MD, Principal Investigator — Ospedale San Luigi Gonzaga, Orbassano, Italy; Arun Rajan, MD., Principal Investigator — National Cancer Institute (NCI); Marina C Garassino, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (6):
- United States (2):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - NIH, Center for Cancer Research, Medical Oncology, Bethesda, Maryland
- France (2):
  - Hopital Larrey, Toulouse
  - Institut de cancerologie Gustave Roussy, Villejuif
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, (MI)
  - Azienda Ospedaliera San Luigi Gonzaga, Orbassano

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 22 February 2010 to 05 April 2016
Groups:
- Milciclib Maleate (PHA-848125AC): 100 and 50 mg Capsule 150 mg/day once daily, for 7 consecutive days (days 1 to 7) followed by 7 days of rest (days 8 to 14) in a 2-week cycle
  Milciclib Maleate: 150 mg/day once daily, for 7 consecutive days (days 1 to 7) followed by 7 days of rest (days 8 to 14) in a 2-week cycle.
  Number of cycles: until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Milciclib Maleate (PHA-848125AC)
Started | 72
Completed | 15
Not Completed | 57
Not completed — Death | 37
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1
Not completed — Sponsor's decision | 15

BASELINE CHARACTERISTICS:
Arm/Group | Milciclib Maleate (PHA-848125AC)
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50
  Black | 2
  Asian | 3
  Not Listed | 10
  Not allowed to ask per local regulation | 6
  Missing | 1
Region of Enrollment [Number; unit: participants]
  United States | 13
  Italy | 36
  France | 23
WHO - Classification [Count of Participants; unit: Participants]
  B3 - Well differantiated thymic carcinoma | 20
  C - Thymic Carcinoma | 52
Tumor extent at study entry [Count of Participants; unit: Participants]
  Locally advanced | 1
  Metastatic | 71
Masaoka clinical staging at study entry [Count of Participants; unit: Participants] — Staging used to evaluate invasiveness of the tumor.
  Participants
    Stage I: grossly and microscopically encapsulated | 0
    Stage II: thymoma invades beyond the capsule | 0
    Stage III: macroscopic invasion neighboring organs | 1
    Stage IV A: pleural or pericardial dissemination | 13
    Stage IVB:hematogeneous or lymphatic dissemination | 51
    Not Listed | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 3 Months
Description: The proportion of successes (i.e. patients alive and progression free at 3 months since treatment start) out of the total number of evaluable patients
Time Frame: 3 months since treatment start
Population: Evaluable patients: population consisting of all treated patients who fulfill the following conditions:
  * histological confirmation of thymic carcinoma by an Independent Review Committee
  * received at least 80% of drug in the first two cycles overall
  * baseline and >/= 1 on treatment tumor assessment or die before tumor re-assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Milciclib Maleate (PHA-848125AC)
Number analyzed (Participants) | 54
Participants
  Success | 24
  Failure | 30
Statistical Analysis 1: Comparison: Milciclib Maleate (PHA-848125AC); H0:p</=17% vs. H1:p>17%, with an interesting PFS-3 rate of 33% or higher; Power=80%; Alpha(1-sided)=5%, 54 evaluable patients are required for a Simon optimal two stage design trial. If at least 4 successes among the first 17 evaluable patients are observed in the 1st stage, patients' enrollment proceed up to the final analysis where at least 14/54 successes (PFS-3 rate ≥ 25.9%) must be required to reject the null hypothesis; Test type: Superiority; p < 0.001, Fisher Exact; Single proportion = 0.44, 95% CI 2-sided [0.31 to 0.59]

2. Secondary Outcome: Confirmed Objective Response Rate (ORR)
Description: Point and 95% confidence interval estimates was calculated for the objective tumor response rate (confirmed CRs or PRs). The determination of antitumor efficacy was based on objective tumor assessments made according to the RECIST guideline (version 1.1) The analysis was performed in the evaluable population.
Time Frame: Assessments were made every 6 weeks from start date until PD to a maximum duration of 242 weeks or until PD.
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Milciclib Maleate (PHA-848125AC)
Number analyzed (Participants) | 54
Percentage of patients | 3.7 [0.45 to 12.75]

3. Secondary Outcome: Disease Control Rate
Description: Point and 95% confidence interval estimates was calculated for the disease control rate (confirmed CRs / PRs and SD>/= 6 weeks). The analysis was performed in the evaluable populations.
Time Frame: Assessments were made every 6 weeks from start date until PD to a maximum duration of 242 weeks or until PD.
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Milciclib Maleate (PHA-848125AC)
Number analyzed (Participants) | 54
Percentage of patients | 75.9 [62.36 to 86.51]

4. Secondary Outcome: Progression-free Survival
Description: The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. In a clinical trial, measuring the progression-free survival is one way to see how well a new treatment works.
Time Frame: Assessments were made every 6 weeks from start date until PD to a maximum duration of 242 weeks or until PD.
Population: Evaluable patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Milciclib Maleate (PHA-848125AC)
Number analyzed (Participants) | 54
Months | 6.83 [4.11 to 8.71]

5. Secondary Outcome: Duration of Response
Description: Assessed in patients achieving a confirmed objective tumor response by RECIST version 1.1 criteria.
Time Frame: Assessments were made every 6 weeks from start date until PD to a maximum duration of 242 weeks or until PD.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Milciclib Maleate (PHA-848125AC): 100 and 50 mg Capsule 150 mg/day once daily, for 7 consecutive days (days 1 to 7) followed by 7 days of rest (days 8 to 14) in a 2-week cycle.
  Milciclib Maleate: 150 mg/day once daily, for 7 consecutive days (days 1 to 7) followed by 7 days of rest (days 8 to 14) in a 2-week cycle.
  Number of cycles: until disease progression or unacceptable toxicity.
Arm/Group | Milciclib Maleate (PHA-848125AC)
Number analyzed (Participants) | 2
Months | 8.41 [6.90 to 9.92]

6. Secondary Outcome: Overall Survival
Description: The length of time from the start of treatment for a disease, such as cancer, to the date in which the patients diagnosed with the disease were still alive.
Time Frame: Every 6 weeks during Follow-Up until PD or new therapy start; every 6 months thereafter, up to 2 years from the last dose of study drug.
Population: Evaluable patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Milciclib Maleate (PHA-848125AC)
Number analyzed (Participants) | 54
Months | 24.18 [16.89 to 36.57]

7. Secondary Outcome: Overall Safety Profile (Adverse Events (NCI CTCAE) and Hematological and Blood Chemistry Parameters)
Description: The adverse events (AEs) were coded with the Medical Dictionary for Regulatory Activities (MedDRA) and their severity graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The following subsets of AEs were considered: serious AEs, AEs with CTCAE grade 3-5, AEs with a relationship to study treatment classified by the Investigator as possible or probable or definite and AEs reported as leading to discontinuation from treatment.
  Laboratory test values were graded according to the NCI CTCAE scale, v3.0, whenever possible. For each laboratory test included in the NCI CTCAE system, the incidence of abnormalities was evaluated by considering the worst occurrence for each patient throughout the whole treatment period.
Time Frame: Adverse events: from date treatment consent signed to 28 days after last dose of study drug; hematology/blood chemistry tests: at baseline and between Day 11-14 of each cycle of a total of 135 two-week cycles.
Population: All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Milciclib Maleate (PHA-848125AC)
Number analyzed (Participants) | 72
Participants
  N° patients with Adverse Events | 72
  N° patients with abnormal Hematology test | 70
  N° patients with abnormal Blood Chemistry test | 70

ADVERSE EVENTS:
Time Frame: Adverse events were reported for patients from consent signed to 28 days after last dose of study drug. Individual patient adverse event reporting ranged from 4.8 weeks to 281.7 weeks with a median of 24.07 weeks.
Arm/Group | Milciclib Maleate (PHA-848125AC)
All-Cause Mortality (participants affected / at risk) | 37/72
Serious Adverse Events (participants affected / at risk) | 22/72
Other Adverse Events (participants affected / at risk) | 72/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milciclib Maleate (PHA-848125AC) (N=72)
Syncope (Nervous system disorders) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Epilepsy NOS (Nervous system disorders) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 1 (2)
Myasthenia gravis (Nervous system disorders) | 1 (1)
Myasthenic syndrome (Nervous system disorders) | 1 (1)
Neuralgia NOS (Nervous system disorders) | 1 (1)
Neurological symptoms (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Sudden death (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Red cell aplasia (Blood and lymphatic system disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 1 (1)
Infection NOS (Infections and infestations) | 1 (1)
Dehydratation (Metabolism and nutrition disorders) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1)
Superior vena caval occclusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milciclib Maleate (PHA-848125AC) (N=72)
Nausea (Gastrointestinal disorders) | 65 (448)
Diarrhoea NOS (Gastrointestinal disorders) | 56 (457)
Vomiting NOS (Gastrointestinal disorders) | 47 (192)
Abdominal pain NOS (Gastrointestinal disorders) | 11 (28)
Abdominal pain upper (Gastrointestinal disorders) | 8 (10)
Constipation (Gastrointestinal disorders) | 8 (15)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 4 (5)
Asthenia (General disorders) | 48 (249)
Chest pain (General disorders) | 14 (30)
Fatigue (General disorders) | 14 (34)
Pyrexia (General disorders) | 10 (13)
Mucosal imflammation (General disorders) | 7 (14)
Oedema peripheral (General disorders) | 5 (10)
Rigors (General disorders) | 5 (5)
Tremor (Nervous system disorders) | 25 (159)
Headache (Nervous system disorders) | 15 (34)
Dysgeusia (Nervous system disorders) | 13 (37)
Dizziness (Nervous system disorders) | 12 (28)
Paraesthesia (Nervous system disorders) | 8 (10)
Dysphonia (Nervous system disorders) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 23 (45)
Hypophosphataemia (Metabolism and nutrition disorders) | 17 (72)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (35)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (28)
Rhinitis NOS (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Alanine aminotransferase increased (Investigations) | 9 (12)
Blood amylase increased (Investigations) | 8 (32)
Lipase increased (Investigations) | 7 (33)
Aspartate aminotransferase increased (Investigations) | 6 (7)
Weight decreased (Investigations) | 5 (5)
Photopsia (Eye disorders) | 7 (14)
Vision blurred (Eye disorders) | 6 (6)
Conjunctivitis (Eye disorders) | 5 (8)
Lacrimation increased (Eye disorders) | 4 (5)
Visual disturbance NOS (Eye disorders) | 4 (5)
Leukopenia NOS (Blood and lymphatic system disorders) | 12 (32)
Neutropenia (Blood and lymphatic system disorders) | 12 (39)
Anaemia NOS (Blood and lymphatic system disorders) | 8 (12)
Rash NOS (Skin and subcutaneous tissue disorders) | 5 (5)
Sweating increased (Skin and subcutaneous tissue disorders) | 4 (7)
Anxiety (Psychiatric disorders) | 6 (12)
Insomnia (Psychiatric disorders) | 6 (12)
Depression (Psychiatric disorders) | 4 (5)
Vertigo (Ear and labyrinth disorders) | 10 (108)
Influenza (Infections and infestations) | 4 (7)
Palpitations (Cardiac disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT01011439/Prot_000.pdf
  • Statistical Analysis Plan: CDKO-125a-006_ALG_V1 (2013-07-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT01011439/SAP_001.pdf
  • Statistical Analysis Plan: CDKO-125a-006_TLG_V1 (2013-07-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT01011439/SAP_002.pdf